CLINICAL TRIAL: NCT04657224
Title: A Phase 1b, Open-Label Study of the Safety, Pharmacokinetics, and Pharmacodynamics of JNJ-64264681 in Combination With JNJ-67856633 in Participants With Non-Hodgkin Lymphoma and Chronic Lymphocytic Leukemia
Brief Title: A Study of JNJ-64264681 and JNJ-67856633 in Participants With Non-Hodgkin Lymphoma and Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108877; 64264681LYM1002 (Other: Janssen Research & Development, LLC); 2020-003149-12 (EudraCT Number); 2024-512687-66-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma, Non-Hodgkin; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — JNJ-64264681

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Dose escalation: JNJ-64264681 and JNJ-67856633 (Experimental): Participants will receive JNJ-64264681 and JNJ-67856633 will be administered together until disease progression, intolerable toxicity, withdrawal of consent, or the investigator.
  Interventions: Drug: JNJ-64264681; Drug: JNJ-67856633
- Part B: Cohort Expansion: JNJ-64264681 and JNJ-67856633 (Experimental): Participants will receive JNJ-64264681 and JNJ-67856633 at the recommended Phase 2 dose (RP2D) determined in Part 1.
  Interventions: Drug: JNJ-64264681; Drug: JNJ-67856633

INTERVENTIONS:
Drug: JNJ-64264681 — JNJ-64264681 capsules will be administered orally.
Drug: JNJ-67856633 — JNJ-67856633 capsules or tablets will be administered orally.

SUMMARY:
The primary purpose of this study is to determine: the recommended Phase 2 doses (RP2Ds) of JNJ-64264681 and JNJ 67856633 when administered together in participants with B cell non-Hodgkin lymphoma (NHL) and chronic lymphocytic leukemia (CLL) (Part A - Dose Escalation); and the safety of the RP2Ds for this combination in different histologies/participant populations (Part B - Cohort Expansion).

DETAILED DESCRIPTION:
Bruton's tyrosine kinase (BTK) is a cytoplasmic tyrosine kinase that plays a critical role in B cell activation via the B cell receptor (BCR) signaling pathway. BTK is important for normal B-cell activation and the pathophysiology of B cell malignancies. A few BTK inhibitors have demonstrated clinical activity in non-Hodgkin lymphoma (NHL) and chronic lymphocytic leukemia (CLL). Non-Hodgkin lymphoma represents a diverse set of diseases, of which more than 60 subtypes have been identified and classified by the world health organization. JNJ-64264681 is a second-generation, orally active, selective, and irreversible covalent inhibitor of BTK and JNJ-67856633 is an orally bioavailable, potent, and selective first in class mucosa-associated lymphoid tissue lymphoma translocation protein 1 (MALT1) inhibitor that binds to an allosteric site on MALT1 with a mixed-type mechanism. JNJ-64264681 and JNJ-67856633 inhibit BTK and MALT1, respectively, and both BTK and MALT1 are involved in transmitting the pro-survival BCR signal. The study will consist of Screening Phase (28 days); Treatment Phase (from Cycle 1 Day 1 up to end of treatment, each cycle is a 21-day cycle) and a Follow-up Phase (from end of treatment visit until lost to follow-up, withdrawal of consent, death, 6 months after start of first subsequent antineoplastic therapy, after the clinical cut off (CCO) date participants will be withdrawn from the study 30 days after the last dose of study drugs were administered). The total study duration is estimated at 2 years and 2 months. Safety assessments will include physical examinations, vital signs, electrocardiograms, clinical safety laboratory assessments, eastern cooperative oncology group performance status, echocardiogram, and adverse events monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1
* Cardiac parameters within the following range: corrected QT interval (QTcF) <= 480 milliseconds
* Participants with B cell non-Hodgkin lymphoma (NHL) must have tumor tissue available at baseline as described in the protocol. This is not required for participants with chronic lymphocytic leukemia (CLL)
* Women of childbearing potential must agree to use a barrier method of contraception; use a highly effective preferably user-independent method of contraception; not to donate eggs (ova, oocytes) or freeze them for future use for the purposes of assisted reproduction during the study; not to plan to become pregnant; and not to breast-feed

Exclusion Criteria:

* Part A and select cohorts in Part B: Prior treatment with JNJ 64264681 or JNJ-67856633. Previously discontinued treatment with a Bruton's tyrosine kinase (BTK) or mucosa-associated lymphoid tissue lymphoma translocation protein (MALT) inhibitor other than JNJ 64264681 or JNJ-67856633 due to participant or doctor choice without evidence of progression or intolerable class-related toxicity will be eligible
* Known (active) central nervous system (CNS) involvement
* Received prior solid organ transplantation
* Participant has known allergies, hypersensitivity, or intolerance to JNJ-64264681 or JNJ 67856633 or excipients
* Toxicities from previous anti-cancer therapies that have not resolved to baseline levels, or to Grade less than (<) 2 (except for alopecia [>=Grade 2], vitiligo [Grade 2] and peripheral neuropathy [Grade 1])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
Part A: Number of Participants with Dose-limiting Toxicity (DLT) | Up to 28 days
  Number of participants with DLT will be assessed. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.
Part A and Part B: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 3 years and 9 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

SECONDARY OUTCOMES:
Plasma Concentrations of JNJ-64264681 and JNJ-67856633 | Up to 3 years and 9 months
  Plasma concentrations of JNJ-64264681 and JNJ-67856633 will be assessed.
Bruton's Tyrosine Kinase (BTK) Occupancy in Peripheral Blood Mononuclear Cell (PBMCs) | Up to 3 years and 9 months
  BTK occupancy will be assessed.
Overall Response Rate (ORR) | Up to 3 years and 9 months
  ORR is defined according to Non-Hodgkin Lymphoma, International Workshop on Chronic Lymphocytic Leukemia (iwCLL); and Response assessment in Waldenström Macroglobulinemia (IWWM).
Time to First Response | Up to 3 years and 9 months
  Time to first response defined for the responders as the time from the date of first dose of study treatment to the date of initial documentation of a first response as defined in the disease-specific response criteria.
Duration of Response | Up to 3 years and 9 months
  DOR will be calculated from the date of initial documentation of a response to the date of first documented evidence of relapse, as defined in the disease-specific response criteria, or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trials, Study Director — Janssen Research & Development, LLC
Locations (28):
- Stony Brook University Medical Center, Stony Brook, New York, United States
- Australia (4):
  - Monash Medical Centre, Clayton
  - Peter MacCallum Cancer Centre, Melbourne
  - Linear Clinical Research Ltd, Nedlands
  - Scientia Clinical Research, Randwick
- Belgium (3):
  - AZ St.-Jan Brugge-Oostende AV, Bruges
  - Universitair Ziekenhuis Gent - UZ GENT, Ghent
  - CHU UCL Namur - Site Godinne, Yvoir
- France (4):
  - CHRU de Lille Hopital Claude Huriez, Lille
  - Chu Hotel Dieu, Nantes
  - Centre hospitalier Lyon-Sud, Pierre-Bénite
  - CHU Bretonneau, Tours
- Arensia Exploratory Medicine, Tbilisi, Georgia
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky MC, Tel Aviv
- Arensia Exploratory Medicine, Chisinau, Moldova
- Academic Medical Center, Amsterdam, Netherlands
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Pratia Onkologia Katowice, Katowice
  - Pratia MCM Krakow, Krakow
  - Centrum Medyczne Pratia Poznan, Skorzewo
- South Korea (3):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (2):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
- Medical Center of Limited Liability Company Arensia Exploratory Medicine, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency